CLINICAL TRIAL: NCT00154440
Title: Treatment of Low-Grade Gastric Non-Hodgkin's Lymphoma of Mucosa-Associated Lymphoid Tissue (MALT) Type Stages IE & II1E (HELYX-Study)
Brief Title: Helicobacter - Lymphoma - Radiation Part I: Eradication, Part II: Radiation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELYX Study
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Lymphoma; Lymphoma, Non-Hodgkin
Keywords: primary gastric MALT lymphoma; Helicobacter pylori; eradication therapy; radiation; marginal zone B-cell lymphoma; Mucosa-associated Lymphoid Tissue; B-cell Non-Hodgkin's Lymphoma of the stomach; primary gastric lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Familial primary gastric lymphoma | interventions — Proton Pump Inhibitors; Clarithromycin; Amoxicillin; Metronidazole; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: proton pump inhibitor
Drug: clarithromycin
Drug: amoxicillin
Drug: metronidazole
Procedure: radiation therapy

SUMMARY:
The first objective of this study is to confirm the results of complete remission of low-grade gastric MALT lymphoma stage IE & II1E after H. pylori eradication on a larger number of patients (HELYX Part I). If there is no response to the antibiotic therapy, the role of radiotherapy on the course of gastric MALT lymphoma will be investigated as a consecutive therapeutic option for patients that are H. pylori- negative, t(11;18)-positive or failure candidates after eradication therapy. Furthermore, the method of radiation, and the radiation dose will be investigated and standardized. HELYX PART II is therefore a randomized equivalent study comparing the standard dose of 36Gy vs. a reduced dose of 25.2Gy locoregional. Additional molecular genetic analysis will be performed to try to understand pathogenetic mechanisms of lymphomagenesis.

DETAILED DESCRIPTION:
Experimental data have extended the knowledge of the mere association of gastric MALT lymphoma and infection with Helicobacter pylori. If we summarise the reports to date on the results of treatment of gastric low-grade MALT lymphoma in an early clinical stage (EI) by H. pylori eradication we find a complete remission figure of 77% in more than 200 patients.

As a therapy with less side effects than radiation, surgery or chemotherapy and as a stomach-conserving treatment, eradication of H. pylori in patients with low-grade gastric MALT lymphoma in stages IE & II1E should be the treatment of the choice within clinical trials since there are no long-term results available thus far. Besides, pretreatment patient selection and careful follow-up with endoscopy, biopsies and clinical staging including endoscopic ultrasonography is necessary. However, a five to ten year-follow-up will be necessary before the definitive value of Helicobacter pylori eradication can be established. Furthermore, since not all patients respond to this therapy research into the pathogenetic mechanisms of lymphomagenesis is inevitable.

Approximately 20% of patients with antigen-positive, primary gastric low-grade MALT lymphoma in stage I will not respond to eradication therapy. Hence, a consecutive salvage therapy other than surgery is much needed. The aim of the second part of this study is to establish radiation therapy as a salvage therapy. Furthermore, the effect of a reduced radiation dose (25.2Gy) compared to the standard dose (36Gy) will be investigated with the aim of non-inferiority of both doses.

ELIGIBILITY:
Inclusion Criteria:

* histologically diagnosed, primary gastric low-grade B-cell MALT lymphoma stages IE or II1E, Helicobacter pylori-positive (in histology, urease test , and serology) for inclusion into HELYX part I
* histologically diagnosed, primary gastric low-grade B-cell MALT lymphoma stages IE or II1E, Helicobacter pylori-negative (in histology, urease test, and serology) for inclusion into HELYX part II
* patients who achieved a study end point of HELYX I: partial remission or no change 12 months after successful antibiotic therapy for inclusion into HELYX part II,
* age > 18 and < 75 years
* Karnofsky-Index > 60%
* sufficient liver function, defined as bilirubin < 34µmol/l
* sufficient renal function, defined as creatinine < 133µmol/l
* written informed consent
* complete clinical tumor staging

Exclusion Criteria:

* primary gastric low-grade MALT lymphoma, stages >II1E or gastric high-grade lymphoma or other lymphoma entities of the stomach e.g. lymphoblastic lymphoma or Burkitt's lymphoma
* age < 18 and > 75 years
* Karnofsky-Index < 60%
* insufficient liver and renal function (see above)
* HIV-infection
* pregnancy or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-11; Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
remission status after eradication therapy 3-monthly
continuous complete remission (CCR) during follow-up
remission status after radiation therapy (36 Gy vs 25.2 Gy)
continuous complete remission after radiation therapy during follow-up

SECONDARY OUTCOMES:
endoscopic controls every 3 months during the first year
endoscopic controls twice yearly in the second year after CR
complete tumor staging once yearly
relapse after therapy after each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morgner-Miehlke, MD, PhD, Principal Investigator — Med. Dept. I, University Hospital, Technical University Dresden
Locations (3):
- Germany (3):
  - Institute for Pathology, Bayreuth, Bavaria
  - Med. Dept. I, Gastroenterology, Dresden, Saxony
  - Dept. for Radiation Therapy & Radiooncology, University Hospital, Germany, Saxony

REFERENCES:
- [Background] Akagi T, Motegi M, Tamura A, Suzuki R, Hosokawa Y, Suzuki H, Ota H, Nakamura S, Morishima Y, Taniwaki M, Seto M. A novel gene, MALT1 at 18q21, is involved in t(11;18) (q21;q21) found in low-grade B-cell lymphoma of mucosa-associated lymphoid tissue. Oncogene. 1999 Oct 14;18(42):5785-94. doi: 10.1038/sj.onc.1203018. PMID 10523859
- [Background] Alpen B, Neubauer A, Dierlamm J, Marynen P, Thiede C, Bayerdorfer E, Stolte M. Translocation t(11;18) absent in early gastric marginal zone B-cell lymphoma of MALT type responding to eradication of Helicobacter pylori infection. Blood. 2000 Jun 15;95(12):4014-5. No abstract available. PMID 10939796
- [Background] Bayerdorffer E, Neubauer A, Rudolph B, Thiede C, Lehn N, Eidt S, Stolte M. Regression of primary gastric lymphoma of mucosa-associated lymphoid tissue type after cure of Helicobacter pylori infection. MALT Lymphoma Study Group. Lancet. 1995 Jun 24;345(8965):1591-4. doi: 10.1016/s0140-6736(95)90113-2. PMID 7783535
- [Background] Hussell T, Isaacson PG, Crabtree JE, Spencer J. The response of cells from low-grade B-cell gastric lymphomas of mucosa-associated lymphoid tissue to Helicobacter pylori. Lancet. 1993 Sep 4;342(8871):571-4. doi: 10.1016/0140-6736(93)91408-e. PMID 8102718
- [Background] Liu H, Ruskon-Fourmestraux A, Lavergne-Slove A, Ye H, Molina T, Bouhnik Y, Hamoudi RA, Diss TC, Dogan A, Megraud F, Rambaud JC, Du MQ, Isaacson PG. Resistance of t(11;18) positive gastric mucosa-associated lymphoid tissue lymphoma to Helicobacter pylori eradication therapy. Lancet. 2001 Jan 6;357(9249):39-40. doi: 10.1016/S0140-6736(00)03571-6. PMID 11197361
- [Background] Neubauer A, Thiede C, Morgner A, Alpen B, Ritter M, Neubauer B, Wundisch T, Ehninger G, Stolte M, Bayerdorffer E. Cure of Helicobacter pylori infection and duration of remission of low-grade gastric mucosa-associated lymphoid tissue lymphoma. J Natl Cancer Inst. 1997 Sep 17;89(18):1350-5. doi: 10.1093/jnci/89.18.1350. PMID 9308704
- [Background] Schechter NR, Portlock CS, Yahalom J. Treatment of mucosa-associated lymphoid tissue lymphoma of the stomach with radiation alone. J Clin Oncol. 1998 May;16(5):1916-21. doi: 10.1200/JCO.1998.16.5.1916. PMID 9586910
- [Background] Thiede C, Morgner A, Alpen B, Wundisch T, Herrmann J, Ritter M, Ehninger G, Stolte M, Bayerdorffer E, Neubauer A. What role does Helicobacter pylori eradication play in gastric MALT and gastric MALT lymphoma? Gastroenterology. 1997 Dec;113(6 Suppl):S61-4. doi: 10.1016/s0016-5085(97)80014-5. PMID 9394762
- [Background] Ruskone-Fourmestraux A, Dragosics B, Morgner A, Wotherspoon A, De Jong D. Paris staging system for primary gastrointestinal lymphomas. Gut. 2003 Jun;52(6):912-3. doi: 10.1136/gut.52.6.912. No abstract available. PMID 12740354
- [Derived] Schmelz R, Miehlke S, Thiede C, Brueckner S, Dawel M, Kuhn M, Ruskone-Formestraux A, Stolte M, Jentsch C, Hampe J, Morgner A. Sequential H. pylori eradication and radiation therapy with reduced dose compared to standard dose for gastric MALT lymphoma stages IE & II1E: a prospective randomized trial. J Gastroenterol. 2019 May;54(5):388-395. doi: 10.1007/s00535-018-1517-4. Epub 2018 Oct 16. PMID 30327875